CLINICAL TRIAL: NCT01140620
Title: Effects of NMDA Receptor Antagonism on Cognitive Processes in Healthy Volunteers and Its Reversal by a Dopamine Antagonist: Comparison to Patients With Schizophrenia
Brief Title: Effects of Ketamine and Risperidone on Cognition
Acronym: Schiz_2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Cardiff University (Other); King's College London (Other); P1vital Limited (Industry)
Responsible Party: Principal Investigator, Bill Deakin, Professor of Psychiatry, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: P1V-SCH-CT02-09
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers; Schizophrenia
Keywords: NMDA receptor antagonism; cognitive processes; healthy volunteers; dopamine antagonist; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine; Risperidone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ketamine and risperidone (Experimental): Oral risperidone pretreatment and intravenous ketamine infusion
  Interventions: Drug: ketamine; Drug: risperidone
- ketamine and placebo (Active Comparator): Oral placebo risperidone pretreatment and intravenous ketamine infusion
  Interventions: Drug: ketamine; Drug: placebo risperidone
- saline and risperidone (Active Comparator): Oral risperidone pretreatment and intravenous saline infusion
  Interventions: Drug: risperidone; Drug: saline
- saline and placebo (Placebo Comparator): Oral placebo risperidone pretreatment and intravenous saline infusion
  Interventions: Drug: saline; Drug: placebo risperidone
- Patients with Schizophrenia (No Intervention): Patients with schizophrenia will not receive study drug and will not undergo randomisation.

INTERVENTIONS:
Drug: ketamine — ketamine infusion to achieve plasma concentrations of 100 ng/mL. Duration approximately 3 hours
  Other Names: ketalar
  Arms: ketamine and placebo; ketamine and risperidone
Drug: risperidone — risperidone (2 mg) capsule. One dosing of 2 mg.
  Other Names: risperdal
  Arms: ketamine and risperidone; saline and risperidone
Drug: saline — saline infusion. Duration approximately 3 hours
  Arms: saline and placebo; saline and risperidone
Drug: placebo risperidone — placebo capsule to match risperidone 2 mg capsule
  Other Names: placebo risperdal
  Arms: ketamine and placebo; saline and placebo

SUMMARY:
The primary objective of this study is:

• To determine the effects of ketamine, which blocks the ion-channel gated by the NMDA receptor, on performance of cognitive tasks and the extent to which these effects can be reversed by the dopamine receptor antagonist, risperidone.

The secondary objectives of this study are:

* To establish whether patients with schizophrenia are able to reliably complete the biomarker test battery and to assess whether their responses are similar to healthy volunteers treated with ketamine.
* To establish a multi-site recruitment and assessment capacity based on shared Standard Operating Procedures across three study centres.

DETAILED DESCRIPTION:
This study is a continuation from a previous study (P1V-SCH-CT01-07). The overall aim of the 2 studies is to identify and validate potential biomarker tasks that may be used to provide early indications into the use of new treatments for schizophrenia. The studies are considering two potential models for schizophrenia in healthy volunteers, the first model looks at high versus average schizotypy, schizotypy being a personality trait. The second model, explored in this study, is a ketamine infusion.

Healthy volunteers will be identified through advertising and will initially be asked to complete an online questionnaire.Suitability for the next stage of the study will be based on the responses to the online questionnaire. Telephone interviews will then be conducted to assess suitability for screening.Screening visits will then be carried out in which a full medical and lab screening is undertaken. participants will also complete a number of psychiatric questionnaires and interviews. If participants remain suitable they will be invited to an assessment day in which they will be randomised to one of four study medication arms. Participants will then complete the biomarker tasks followed by questionnaires, rating scales and interviews. Patients with schizophrenia will form the 5th study arm and will not receive medication. They will complete the biomarkers in the same way as healthy volunteers.87 participants are planned, 72 healthy volunteers, 15 patients with schizophrenia.

This study does not test any investigational medicinal product (IMP) so any ethical issues that are associated with introducing a participant to a study drug are not applicable in this study.

Ketamine is already a widely used anaesthetic agent but when given at sub-anaesthetic doses is a useful tool for modelling schizophrenia psychosis.

The current study aims to assess the sensitivity of a battery of biomarker tasks (biomarkers are measures of processes that go wrong in illnesses and that contribute to symptoms) to the cognitive deficits induced by ketamine.

It may in future be possible to evaluate the effects of novel treatment for schizophrenia in healthy volunteers using this model, which would then potentially provide a rapid indication of the potential efficacy of candidate compounds at an early phase of drug development .

The study will provide information about the sensitivity of the biomarker tasks in detecting the effects of the pharmacological treatments for schizophrenia in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

5.2.1 General inclusion criteria (healthy and schizophrenia groups)

* Male or female aged 18 to 45 years
* Fluent English speakers, preferably with English as first language.
* Normotensive with sitting (5 minutes) blood pressure of 100 to 140 mmHg systolic, and 60 to 90 mmHg diastolic.
* Negative alcohol breath test.
* Negative urine drug screen.
* Participant must have consumed only their normal intake of coffee or tea on the morning of the assessment day and not consumed any other beverages containing caffeine for 2 hours prior to the assessment visit.
* Willing to follow the protocol prohibitions and restrictions .
* Participant must have signed the informed consent form.
* Those participants willing to participate in the pharmacogenomic components of the study must have signed the appropriate informed consent form.

5.2.2 Inclusion criteria applicable to healthy volunteers only

* SPQ score of 21 to 36.
* BMI of 18 to 30 kg/m².
* Non-smoker or light smoker (less than 5 cigarettes per day).
* Has not smoked in the 2 hours prior to the assessment visit.
* Females should be surgically sterile or abstinent or practising an effective method of birth control; they should have a negative urine pregnancy test.
* Healthy at screening and assessment visits as determined by the study physician, based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs, 12-lead ECG and pre-study psychological tests.

5.2.3 Inclusion criteria applicable to participants with schizophrenia only

* Documented history of a diagnosis of schizophrenia as confirmed by GP or psychiatrist or by previous research diagnostic interview.
* Confirmation of diagnosis of schizophrenia, based on the MINI structured clinical interview, carried out by the study physician.
* In good physical health at screening and assessment visits as determined by the study physician, based on a medical evaluation including medical history, physical examination, laboratory tests and vital signs1.

Exclusion Criteria:

5.3.1 General exclusion criteria (healthy and schizophrenia groups)

* History of alcohol or substance dependence.
* Consumption of large amounts of caffeinated drinks.
* Have received over-the-counter medicine within 48 hours prior to assessment visit (apart from paracetamol) unless it will not interfere with the study procedures or compromise safety.
* History of, or current condition of, migraine headaches.
* Significant hearing impairment which in the opinion of the Investigator may interfere with the performance of the psychological test battery.
* Significant visual impairment or history of ocular treatment or ongoing condition which may interfere with the performance of the psychological test battery.
* Participated in a trial with any drug within 84 days of assessment visit.
* Unable or unwilling to comply with study procedures.

5.3.2 Exclusion criteria applicable to healthy volunteers only

* Known or suspected hypersensitivity or intolerance to risperidone or any of their excipients.
* Known or suspected hypersensitivity or intolerance to ketamine or any previous adverse reaction to anaesthesia.
* If female: are pregnant or are trying to get pregnant or are currently breast feeding.
* Relevant history, or presence upon clinical examination, of cardiac, ophthalmologic, gastro-intestinal, hepatic, or renal disease or other condition known to increase risk of side effects.
* History or presence of neurological or psychiatric conditions.
* Have received prescribed medication within 14 days prior to assessment visit (apart from the contraceptive pill) unless it will not interfere with the study procedures or compromise safety.

5.3.3 Exclusion criteria applicable to participants with schizophrenia only

* Changes to antipsychotic medications within 30 days of assessment visit.
* Admission to hospital, involvement with the home treatment team for psychiatric reasons or documented relapse of psychiatric symptoms within last 3 months.
* History or presence of psychiatric or neurological conditions other than schizophrenia, major depression and generalised anxiety disorder.
* Current extra-pyramidal symptoms and/or adverse effects from antipsychotic medications that, in the opinion of the study physician, will interfere with completion of the study tasks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Biconditional learning task | 6 months
  Accuracy (% correct) for simple and biconditional learning trials, averaged over 8 blocks
Eye movement task | 6 months
  1. Antisaccade error rate.
  2. Antisaccade correction rate.
  3. Antisaccade latency.
  4. Antisaccade amplitude gain.
  5. Antisaccade peak velocity.
  6. Prosaccade error rate.
  7. Prosaccade correction rate.
  8. Prosaccade latency.
  9. Prosaccade amplitude gain.
  10. Prosaccade peak velocity.
  11. Smooth pursuit gain at three different target speeds.
  12. Smooth pursuit saccadic frequency at three different target speeds.
Salience Attribution task | 6 months
  1. Implicit aberrant salience (ms).
  2. i. Overall reaction time
  b.ii. Implicit adaptive salience (ms).
  c. Explicit adaptive salience (mm).
  d. Explicit aberrant salience (mm).
  e. Commission errors.
  f. Omission errors.
Signal detection task | 6 months
  1. d׳ value
  2. Hits, when participants respond positively and a voice is present.
  3. False alarm rate.
  4. β value.
N-Back | 6 months
  1. Correct responses across three levels of difficulty.
  2. Percentage of overall responses that was correct.
  3. Errors of omission.
  4. Errors of commission.
Spatial working memory | 6 months
  1. Between search error rate - errors due to a participant returning to a treasure chest which had previously contained some treasure on an earlier trial within the same block.
  2. Within search error rate - errors due to a participant returning to the same treasure chest more than once within a trial.
  3. Average time to complete each difficulty level
Verbal Fluency | 6 months
  1. Number of words generated.
  2. Number of repetition errors: When the same word is repeated more than once within the letter or category.
  3. Number of set loss errors: These are: i.) Words that start with a letter which do not fit the trial; ii.) Words which are names of people or places or numbers; iii.) Grammatical variants of an already stated word; and iv.) Non-words.
Event-related potentials (Manchester EEG pilot study only) | 6 months
  1. Amplitude and latencies of the positive peak in the 80-160 ms range (P1) and the negative peak in the 160 - 250 ms range (N1) for the Kanitsa and non-Kanitsa conditions.
  2. Evoked gamma (30-100 Hz) and beta (14-30 Hz) oscillations in the 30 - 350 ms range to the Kanitsa condition.
  3. Evoked alpha (8-12 Hz) and theta (4-8 Hz) oscillations in the 30-500 ms range to both conditions.
  4. Coherence within and between frontal and occipital electrodes in the 100 - 400 ms range
Questionnaires and assessment scale scores | 6 months
  1. CADSS.
  2. BPRS.
  3. Effects of Drug Rating Scale.

SECONDARY OUTCOMES:
Pharmacogenomic analysis | 12 months
  An exploratory genetic analysis aiming to correlate any genetic polymorphisms associated with schizotypy, schizophrenia or brain development with study outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Bill Deakin, Principal Investigator — University of Manchester
Locations (3):
- United Kingdom (3):
  - Institute of Psychiatry, King's College London, London, Greater London
  - University of Manchester (Dept of Neuropyschiatry), Manchester, Manchester
  - School of Psychology, University of Cardiff, Cardiff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website — http://www.p1vital.com